CLINICAL TRIAL: NCT00335751
Title: Glucose Metabolic Response by PET/CT to Sarcoma Treatments
Brief Title: PET Scan Combined With CT Scan in Evaluating Treatment Response in Patients Undergoing Treatment for Bone Cancer or Soft Tissue Sarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000480348; UCLA-0508095-01
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2016-01

CONDITIONS: Sarcoma
Keywords: recurrent adult soft tissue sarcoma; stage I adult soft tissue sarcoma; localized osteosarcoma; metastatic osteosarcoma; recurrent osteosarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- positron emission tomography computed tomography (PET/CT) (Experimental): The first PET/CT scan will be performed as part of clinical evaluation of sarcoma; The second PET/CT scan will be performed 6 weeks after the start of chemotherapy treatment OR 6 weeks after the end of radiation therapy, to monitor response of sarcoma to treatment.
  Interventions: Procedure: positron emission tomography computed tomography (PET/CT)

INTERVENTIONS:
Procedure: positron emission tomography computed tomography (PET/CT) — The first PET/CT scan will be performed as part of clinical evaluation of sarcoma; The second PET/CT scan will be performed 6 weeks after the start of chemotherapy treatment OR 6 weeks after the end of radiation therapy, to monitor response of sarcoma to treatment.

SUMMARY:
RATIONALE: Diagnostic procedures, such as PET scan and CT scan, may help doctors determine the extent of cancer and predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This clinical trial is studying how well PET scan combined with CT scan evaluates treatment response in patients undergoing treatment for bone cancer or soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether an FDA-approved device that combines fludeoxyglucose ^18F positron-emission tomography (FDG-PET) and CT scanning (FDG-PET/CT) can accurately locate and determine the extent of disease in patients who are undergoing treatment for bone or soft tissue sarcoma.
* Determine whether FDG-PET/CT scanning is effective in evaluating the response of sarcoma to treatment.
* Determine whether the new FDG-PET/CT device improves the ability to evaluate treatment response early and accurately.
* Correlate changes in glucose metabolic activity early and late after treatment with overall and progression-free survival.
* Correlate changes in glucose metabolic activity early and late after treatment with degree of tumor necrosis at the time of surgery.

OUTLINE: This is a prospective, pilot study. Patients are stratified according to disease (high-grade soft tissue sarcoma vs low-grade soft tissue sarcoma vs osteosarcoma).

Patients undergo fludeoxyglucose ^18F positron-emission tomography (FDG-PET)/CT scanning at baseline and then within 2 weeks and 12 weeks after the start of treatment (total of 3 scans).

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed bone or soft tissue sarcoma
* Scheduled to undergo treatment (i.e., chemotherapy and/or radiotherapy) for sarcoma
* Negative pregnancy test
* Fertile patients must use effective contraception
* Not claustrophobic
* Able to lie supine for 1 hour
* Patients with diabetes mellitus allowed provided serum glucose levels ≤ 200 mg/dL

Exclusion Criteria:

* pregnant
* other malignancies within the past 5 years (except completely resected cervical or nonmelanoma skin cancer) unless the malignancy was curatively treated and is at low risk for recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Determine whether device that combines fludeoxyglucose ^18F positron-emission tomography (FDG-PET) and CT scanning (FDG-PET/CT) can accurately locate and determine disease in patients who are undergoing treatment for bone or soft tissue sarcoma. | 6 months

SECONDARY OUTCOMES:
•Determine whether FDG-PET/CT scanning is effective in evaluating the response of sarcoma to treatment. | 6 months
•Determine whether the new FDG-PET/CT device improves the ability to evaluate treatment response early and accurately. | 6 months
•Correlate changes in glucose metabolic activity early and late after treatment with overall and progression-free survival. | 6 months
•Correlate changes in glucose metabolic activity early and late after treatment with degree of tumor necrosis at the time of surgery. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No